CLINICAL TRIAL: NCT02387151
Title: Safety of Allogeneic Bone Marrow Derived Mesenchymal Stromal Cell Therapy in Renal Transplant Recipients
Brief Title: Allogeneic Mesenchymal Stromal Cell Therapy in Renal Transplant Recipients
Acronym: Neptune
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, M.E. J. Reinders, MD/PhD, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL4724400013; 2013-005407-14 (EudraCT Number)
Record Dates: First submitted 2015-03-03; First posted 2015-03-12 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Rejection; Graft Loss
Keywords: Mesenchymal Stromal Cells; Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mesenchymal stromal cells (Experimental): allogeneic mesenchymal stromal cell infusion
  Interventions: Drug: mesenchymal stromal cells

INTERVENTIONS:
Drug: mesenchymal stromal cells — 2 doses of 1-2x10^6 allogeneic bone marrow derives MSCs IV per/kg body weight at weeks 25 and 26 after transplantation
  Other Names: MSC; bone marrow derived mesenchymal stromal cells

SUMMARY:
This study will test whether selected allogeneic bone marrow derived MSCs are safe by assessing the composite end point Biopsy Proven Acute Rejection (BPAR)/ graft loss at 12 months.

DETAILED DESCRIPTION:
Kidney transplantation has improved survival and quality of life for patients with end-stage renal disease. However, despite advances in immunosuppressive therapy, long-term allograft survival outcomes have not improved over the last decade.

A promising novel therapeutic immunosuppressive option in the treatment of renal recipients with a profound effect on the fibrosis reaction is the clinical application of mesenchymal stromal cells (MSCs). Allogeneic MSCs offer the advantage of availability for clinical use without the delay required for expansion.

Although it is believed that allo MSCs are immune privileged, they could possibly elicit an anti-donor immune response, which may increase the incidence of rejection/ graft loss and impact the allograft survival on the long term. These safety issues should be studied before further studies are planned with allogeneic MSCs in the transplant setting.

MSCs are infused at a time point when immune suppression is lowered and the kidney is at increased risk for developing immune mediated injury. In addition, a large amount of the kidneys already has signs of fibrosis at this time point and MSCs might reduce the fibrosis which so importantly affects long term survival. MSCs will have no Human Leucocyte Antigen (HLA) sharing with the mismatches of the donor and the recipient should have no antibodies directed to the MSCs to reduce the anti-donor immune respons risk.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to participate in the study, must be able to give informed consent and the consent must be obtained prior to any study procedure.
* Recipients of a first kidney graft from a living-unrelated or non-HLA identical living related donor.
* Panel Reactive Antibodies (PRA) ≤ 50%.
* Patients must be able to adhere to the study visit schedule and protocol requirements.
* If female and of child-bearing age, subject must be non-pregnant, non-breastfeeding, and use adequate contraception.

Exclusion Criteria:

* Double organ transplant recipient.
* Biopsy proven acute rejection (according to the Banff criteria) in the 4 weeks before MSC infusion.
* Patients with evidence of active infection or abscesses (with the exception of an uncomplicated urinary tract infection) before MSC infusion.
* Patients suffering from hepatic failure.
* Patients suffering from an active autoimmune disease.
* A psychiatric, addictive or any disorder that compromises ability to give truly informed consent for participation in this study.
* Use of any investigational drug after transplantation.
* Documented HIV infection, active hepatitis B, hepatitis C or tuberculosis according to current transplantation inclusion criteria.
* Subjects who currently an active opportunistic infection at the time of MSC infusion (e.g., herpes zoster [shingles], cytomegalovirus (CMV), Pneumocystis carinii (PCP), aspergillosis, histoplasmosis, or mycobacteria other than tuberculosis, BK) after transplantation.
* Malignancy (including lymphoproliferative disease) within the past 2-5 years (except for squamous or basal cell carcinoma of the skin that has been treated with no evidence of recurrence) according to current transplantation inclusion criteria
* Known recent substance abuse (drug or alcohol).
* Patients who are recipients of ABO incompatible transplants.
* Patients with severe total hypercholesterolemia (>7.5 mmol/L) or total hypertriglyceridemia (>5.6 mmol/L) (patients on lipid lowering treatment with controlled hyperlipidemia are acceptable).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
biopsy proven acute rejection / graft loss | 12 months after transplantation

SECONDARY OUTCOMES:
Comparison of fibrosis by quantitative Sirius Red scoring | Before MSC infusion (week 24 after transplantation) and 6 months after MSC infusion (week 52 after transplantation)
Serious adverse events | 12 months after transplantation
Renal function measured by cGFR (MDRD formula) and iohexol clearance | week 24 after transplantation (before MSC infusion) and 52 after transplantation
CMV, BK infection (viremia, disease and syndrome; and subtypes of BK viremia) and other opportunistic infections | from baseline up to 26 weeks after MSC treatment
Development of de novo donor specific antibodies (DSA) and immunological responses | at baseline, week 24 after transplantation (before MSC treatment) up to week 26 after MSC treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marlies EJ Reinders, MD/PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Reinders ME, Dreyer GJ, Bank JR, Roelofs H, Heidt S, Roelen DL, Zandvliet ML, Huurman VA, Fibbe WE, van Kooten C, Claas FH, Rabelink TJ, de Fijter JW. Safety of allogeneic bone marrow derived mesenchymal stromal cell therapy in renal transplant recipients: the neptune study. J Transl Med. 2015 Nov 4;13:344. doi: 10.1186/s12967-015-0700-0. PMID 26537851